CLINICAL TRIAL: NCT06228599
Title: Molecular Profile-related Individualized Targeted Therapy in Resected Pancreatic Cancer With High-Risk of Cancer Recurrence
Acronym: PROTECT-PANC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mandana Kamgar, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00049951
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pancreas Cancer
Keywords: pancreatic cancer; molecular profile; targeted therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Molecular Tumor Board (MTB)-recommended matched therapy (Experimental): The MTB, a multidisciplinary group composed of medical oncologists (including those with expertise in precision oncology), surgical oncologists, and a pathologist, convenes periodically to discuss and recommend an individualized treatment plan that targets specific molecular alterations (e.g., genomic mutations) found in the patient's cancer while considering patient clinical and laboratory factors.
  Interventions: Other: Treatment Plan

INTERVENTIONS:
Other: Treatment Plan — A matched treatment regimen will be administered for approximately 12 weeks based on recommendations made by the MTB.

SUMMARY:
This is a prospective, open-label therapeutic interventional investigation designed to interrogate the efficacy and safety of individualized matched therapies in patients with pancreatic cancer at high risk of disease recurrence post-surgery.

DETAILED DESCRIPTION:
This is a prospective, open-label, therapeutic interventional investigation designed to interrogate the efficacy and safety of personalized matched therapy in pancreatic cancer patients who have completed all intended multimodal therapy, including resection of the pancreatic cancer tumor. Potential participants must have their tumor tissue or blood molecularly profiled with the results discussed by the Molecular Tumor Board, whether convened in person, virtually (e.g., WebEx), or in an electronic forum (e.g., email). Only those patients who agree to receive the Molecular Tumor Board-recommended matched therapy (i.e., study treatment) will be eligible and enrolled on the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Pathologically confirmed pancreatic cancer (excluding neuroendocrine histology).
3. Pancreatic tumor is surgically removed and

   1. patient has received multimodal therapy (neoadjuvant, sandwich or adjuvant chemotherapy ± radiation) or
   2. patient is ineligible for or refuses multimodal therapy.
4. Patient has one of the following:

   1. Post-surgical cancer antigen (CA) 19-9 elevation (> 35 U/mL at least 6 weeks post-surgical resection) in the setting of bilirubin < 2 mg/dL (unless bilirubin elevation is consistent with Gilbert's syndrome) OR
   2. High-risk pathological features, defined as positive surgical margin or lymph node involvement in cancer.
5. Patient has no definitive measurable disease recurrence or metastatic disease at the time of first post-surgical imaging (in those with high-risk pathological features) or within four weeks of elevated CA 19-9 value as evidenced by appropriate imaging.
6. Laboratory values:

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 109/L.
   2. Platelet count ≥ 75,000/mm^3 (125 × 109/L).
   3. Hemoglobin (Hgb) ≥ 8 g/dL.
   4. aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT), alanine transaminase (ALT) serum glutamate-pyruvate transaminase (SGPT) ≤ 5 × upper limit of normal range (ULN).
7. Eastern Cooperative Oncology Group (ECOG) Performance Status < 3.
8. At the time of treatment, patient should be off other anti-tumor agents for at least five half-lives of the agent or three weeks from the last day of treatment, whichever is shorter.
9. Able to swallow and retain oral medication, if needed.
10. Pregnancy It is not known what effects matched therapy has on human pregnancy or development of the embryo or fetus. Therefore, female subjects participating in this study should avoid becoming pregnant, and male subjects should avoid impregnating a female partner. Nonsterilized female subjects of reproductive age and male subjects should use effective methods of contraception through defined periods during and after study treatment as specified below.

    Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
    * Not a female of childbearing potential (FCBP), defined as all female patients that were not in post-menopause for at least one year or are surgically sterile, OR
    * An FCBP must have a negative serum pregnancy test and agree to use at least one form of pregnancy prevention during the study for at least one month after treatment discontinuation unless otherwise noted by the agent(s) USPI, which the FCBP must follow.

    Male participants: A male participant, even if surgically sterilized (i.e., status post vasectomy), must use a form of barrier pregnancy prevention approved by the investigator or treating physician during the study and for at least one month after treatment discontinuation and refrain from donating sperm during this period unless otherwise noted by the agent(s) USPI, which the male participant must follow.
11. Patient must be presented at the Molecular Tumor Board (MTB) and agree to receive the MTB-recommended therapy.
12. Ability to understand a written informed consent document, and the willingness to sign it.

    1. Patients presented at the MTB prior to signing consent are eligible to be on study. Patients do not need to be presented again at the MTB prior to starting therapy on trial unless six months elapse between consent and start of study treatment.

Exclusion Criteria:

A potential study subject who meets any of the following exclusion criteria is ineligible to participate in the study.

1. CA 19-9 non-producers, unless high-risk pathological features present.
2. Receiving concomitant investigational agent(s) for pancreatic ductal adenocarcinoma (PDAC).
3. Radiographic evidence of metastatic disease.
4. Inability to ingest study drugs by mouth.
5. Diarrheal bowel movements > 6 per day postoperatively on maximal medical therapy.
6. Patient has active, untreated, or uncontrolled bacterial, viral, or fungal infection(s) requiring systemic intravenous therapy.
7. Patient has undergone or planned major surgery other than diagnostic surgery (i.e., surgery done to obtain a biopsy for diagnosis without removal of an organ) within four weeks prior to Day 1 of study therapy.
8. Patient has a history of allergy or hypersensitivity to the study drug(s) or any of the excipients.
9. Uncontrolled concurrent illness, including, but not limited to, unstable angina pectoris, uncontrolled and clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Is pregnant or breastfeeding or any patient with childbearing potential not using adequate pregnancy prevention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | Six months
  The number of subjects exhibiting disease-free survival at six months. Disease-free survival is defined as the time from study therapy initiation until disease recurrence or death from any cause.
Adverse Events | Up to 12 months
  The number of clinically relevant Grade 3 to 4 adverse events and serious adverse events that are at least possibly related to the study therapy per investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Kamgar, MD, MPH, Principal Investigator — Medical College of Wisconsin; Razelle Kurzrock, MD, Principal Investigator — Medical College of Wisconsin; Douglas Evans, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No